CLINICAL TRIAL: NCT03830294
Title: Physical and Psychological Effects of Different Temperature-controlled Breast Prostheses on Patients With Breast Cancer During Rehabilitation: a Randomized Controlled Study
Brief Title: Physical and Psychological Effects of Different Temperature-controlled Breast Prostheses on Patients With Breast Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhenqi Lu, Director of Nusing Administration, Fudan University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB1403133-2
Record Dates: First submitted 2019-01-25; First posted 2019-02-05 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: External Breast Prostheses
Keywords: breast prostheses, physical, psychological, breast cancer,
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Self-adhesive Group (Experimental): The participants used the adhesive breast prosthesis that adheres to the skin.
  Interventions: Other: different temperature-controlled breast prostheses
- Conventional Group (Active Comparator): The participants used the conventional breast prosthesis that was placed inside a bra and did not directly adhere to the skin.
  Interventions: Other: different temperature-controlled breast prostheses

INTERVENTIONS:
Other: different temperature-controlled breast prostheses — Two types of temperature-controlled breast prostheses were applied to patients in each group

SUMMARY:
Breast loss causes negative influence on women physically, psychologically and socially. Breast prosthesis can improve patient's figure externally, increase self-confidence, thus improving quality of life. The objective was to understand the knowledge regarding breast prostheses in breast cancer patients, evaluate the quality of life of patients wearing different types of breast prostheses and to compare the physical and psychological effects of different temperature-controlled breast prostheses on patients. The investigators designed a randomized control study in one cancer center in Shanghai. In the first 6 weeks of the study, self-adhesive breast prostheses and conventional breast prostheses were used in the intervention and control group, respectively. In the later 6 weeks, the breast prostheses used were switched into another kind. Several dimensional parameters were examined by different questionnaires at the end of both 6th and 12th week including scars and skin, survey of breast prosthesis knowledge, survey assessing the comfort and practicality of breast prostheses, quality of life instruments for cancer patients and body image scale. The investigators expected that women would be satisfied with the temperature-controlled breast prosthesis and were more willing to choose self-adhesive breast prostheses.

DETAILED DESCRIPTION:
Breast loss causes negative influence on women physically, psychologically and socially. Breast prosthesis can improve patient's figure externally, increase self-confidence, thus improving quality of life. Prospective study of different breast prostheses has not yet been performed in China. The objective was to understand the knowledge regarding breast prostheses in breast cancer patients, evaluate the quality of life of patients wearing different types of breast prostheses and to compare the physical and psychological effects of different temperature-controlled breast prostheses on patients. The investigators designed a randomized control study in one cancer center in Shanghai. Eligible participants were randomized into either intervention or control group. In the first 6 weeks of the study, self-adhesive breast prostheses and conventional breast prostheses were used in the intervention and control group, respectively. In the later 6 weeks, the breast prostheses used were switched into another kind. Several dimensional parameters were examined by different questionnaires at the end of both 6th and 12th week including scars and skin, survey of breast prosthesis knowledge, survey assessing the comfort and practicality of breast prostheses, quality of life instruments for cancer patients and body image scale. The investigators expected that women would be satisfied with the temperature-controlled breast prosthesis and were more willing to choose self-adhesive breast prostheses.

ELIGIBILITY:
Inclusion Criteria:

* undergoing unilateral mastectomy due to breast cancer confirmed by histological examination
* had undergone mastectomy at least six months prior to the start of the study or patients who completed radiation therapy at least two months prior
* without evidence of postoperative relapse
* wearing conventional (non-adhesive) breast prostheses
* without abnormal skin or skin lesions
* patients without progressive lymphedema;
* interested in conventional and self-adhesive breast prostheses.

Exclusion Criteria:

* with incomplete healing of their surgical wounds
* undergoing chemoradiotherapy or who received chemoradiotherapy less than two months prior to the beginning of the study
* with skin conditions that do not meet the requirements
* whose remaining breast is not within the study's size range
* with significant life changes during the study, including divorce, unemployment or depression; 6) relapsed during the observation period
* had a reaction to the first skin test and who were not able to receive the second skin test.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-10-10 (Actual); Primary Completion 2017-05-31 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Participants' skin condition | 12 weeks
  Scars and skin conditions: these examinations were performed by the same investigator.
Participants' knowledge with regard to the breast prosthesis | 12 weeks
  A self-designed questionnaire covering a total of 11 items was used, including sources the patients used to obtain information on breast prostheses, reasons for choosing the breast prosthesis, its type and price, and the patient's feelings about wearing their breast prosthesis.
Participants' feeling of the comfort and practicality of breast prostheses | 12 weeks
  A self-designed questionnaire covering a total of 10 items regarding the breast prostheses was used, including skin adhesion, practicality in daily life, maintainability, comfort, natural fit, contact, safety, and effects on the shoulder and back
Measurement of Quality of life of the participants | 12 weeks
  We use breast cancer (QLICP-BR) to measure patients' quality of life.the QLICP-BR selected the following 37 items: 6 items in physical functional dimensions (PH), 12 items in psychological functional dimensions (PS), 8 items in symptoms and side effects dimensions (ST), 10 items in social functional dimensions (SOs) and 1 item in overall health condition.
Measurement of Body Image of the participants | 12 weeks
  The Body Image Scale (BIS) is a self-assessment scale designed to assess cancer patients' perceptions of their appearance and identify any changes to those perceptions resulting from a disease or a treatment.

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] 1.Huang ZZ, Chen WQ, Wu CX, et al. Incidence and mortality of female breast cancer in China--- a report from 32 Chinese cancer registries, 2003-2007. Tumor, 2012, 32(6):435-439. 2.Li N, Zheng RS, Zhang SW, et al. Analysis and prediction of breast cancer incidence trend in China. Chinese Journal of Preventive Medicine, 2012, 8(46):703-707. 3.Huang ZZ, Chen WQ, Wu CX, et al. The trends of female breast cancer incidence and mortality in Beijing, Shanghai, Linzhou and Qidong in China. Tumor, 2012, 32(8): 605-608. 4.Li MF, Wang XH, Zhao XY. Research of breast cancer incidence. Journal of China Traditional Chinese Medicine Information, 2011, 15(3): 76. 5.Chen W, Wang CS, Zhang W. Comparison of breast-conserving therapy and mastectomy. Chinese Primary Medicine, 2013,2(20):255-257. 6.Zhang BN, Yu ZH. Key problems in breast-conserving surgeries. Chinese Journal of Oncology, 2001,23(6):523-524. 7.Zhang BN, Zhang B, Tang ZH, et al. 10-year changes and development of surgical treatment for breast cancer in China. Chinese Journal of Oncology, 2012,8(34): 582-587. 8.Zhang YS, Liu YJ. A review for the surgical management of breast cancer and the latest developments. Modern Oncology, 2015,5(23):719-722. 9.Song YL, Zhang KM. Development of psychological nursing in postoperative breast cancer patients who lost their breasts. Medical Equipment, 2015,2(28):125-126. 10.Sun LQ. Cognitive study on prostheses wearing in postoperative breast cancer patients who lost their breasts. Journal of Qilu Nursing, 2010,16(21):48-49. 11.Xie SH. Physical and psychological influence of breast loss on postoperative breast cancer patients and nursing strategy. Chinese General Practice Nursing, 2014,12(4):351-352. 12.Ding ZY. Perioperative nursing of breast cancer patients who undergone DIEP. Nursing Journal of Chinese People's Liberation Army, 2006,12(24):67-68. 13.Cao RJ. Investigation of sexual status of patients who undergone mastectomy. Today Nurse, 2011(6):114-116. 14.Ren HL, Jia XJ, Wang Q. Correlation between postoperative self-image and coping style of patients with breast cancer. Chinese Journal of Modern Nursing, 2014,20(11):1274-1277. 15.Li R. Effective analysis of different surgical treatments in early-stage breast cancer. Chinese Youjiang Medical Journal, 2013,41(1):4-6. 16.Zhang HX. Analysis of influential factors on quality of life of patients with breast cancer. Nursing Journal of Chinese People's Liberation Army, 2007,24(3):45-46. 17.Huang LP, Xiong BQ. Application of high quality nursing on prostheses wearing in postoperative patients with breast cancer. Journal of Yangtze University(Natural Science Edition), 2013,10(6):42-43. 18.Gallagher P, Buckmaster A, O'Carroll S, et al. Experiences in the provision, fitting and supply of external breast prostheses: findings from a national survey. European Journal of Cancer Care,2009,6(18):556-568. 19.Thijs-Boer FM, Thijs JT, Van HB. Conventional or adhesive external breast prosthesis? A prospective study of the patients' preference after mastectomy. Cancer Nurs,2001,3(24):227-230. 20.Kubon TM, McClennen J, MI Fitch, et al. A mixed-methods cohort study to determine perceived patient benefit in providing custom breast prostheses. Current Oncology, 2012, 2(19):43-52.